CLINICAL TRIAL: NCT02741115
Title: Fontan Udenafil Exercise Longitudinal Assessment Trial (FUEL)
Brief Title: Fontan Udenafil Exercise Longitudinal Assessment Trial
Acronym: FUEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mezzion Pharma Co. Ltd (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHN-Udenafil-02; U01HL068270 (NIH)
Record Dates: First submitted 2016-04-10; First posted 2016-04-18 (Estimated); Results first posted 2025-05-21 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Single Ventricle Heart Disease
Keywords: Fontan; Maximal Oxygen Consumption; Vascular Function; EndoPAT; Myocardial Performance
MeSH Terms: interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug (Experimental): Udenafil. One tablet twice daily for 26 weeks
  Interventions: Drug: Udenafil
- Placebo (Experimental): Placebo. One tablet twice daily for 26 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Udenafil — Active drug
  Arms: Drug
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the clinical efficacy and safety of udenafil, an orally administered, potent and selective inhibitor of PDE5, versus placebo for the treatment of adolescent subjects who have undergone the Fontan procedure.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, efficacy trial of the effects of udenafil vs. placebo on the background of standard therapy on maximal VO2 (ml/kg/min) from baseline to six months in adolescent survivors of the Fontan procedure. . The target sample size is 400 subjects (200 per group).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females with Fontan physiology who are 12 to less than 19 years of age at enrollment.
2. Participant consent or parental/guardian consent and participant assent
3. Participant fluency in primary language of country in which study is being conducted

Exclusion Criteria:

1. Weight < 40 kg
2. Height < 132 cm.
3. Hospitalization for acute decompensated heart failure within the last 12 months.
4. Current intravenous inotropic drugs.
5. Undergoing evaluation for heart transplantation or listed for transplantation.
6. Diagnosis of active protein losing enteropathy or plastic bronchitis within the last 3 years, or a history of liver cirrhosis.
7. Known Fontan baffle obstruction, branch pulmonary artery stenosis, or pulmonary vein stenosis resulting in a mean gradient of > 4 mmHg between the regions proximal and distal to the obstruction as measured by either catheterization or echocardiography, obtained prior to screening for the trial.
8. Single lung physiology with greater than 80% flow to one lung.
9. VO2 less than 50%
10. Severe ventricular dysfunction assessed qualitatively by clinical echocardiography within six months prior to enrollment.
11. Severe valvar regurgitation, ventricular outflow obstruction, or aortic arch obstruction assessed by clinical echocardiography within six months prior to enrollment.
12. Significant renal (serum creatinine > 2.0), hepatic (serum AST and/or ALT > 3 times upper limit of normal), gastrointestinal or biliary disorders that could impair absorption, metabolism or excretion of orally administered medications, based on laboratory assessment six weeks prior to screening for the trial.
13. Inability to complete exercise testing at baseline screening.
14. History of PDE-5 inhibitor use within 3 months before study onset.
15. History of any other medication for treatment of pulmonary hypertension within 3 months before study onset.
16. Known intolerance to oral udenafil.
17. Frequent use of medications or other substances that inhibit or induce CYP3A4.
18. Current use of alpha-blockers or nitrates.
19. Ongoing or planned participation in another research protocol that would either prevent successful completion of planned study testing or invalidate its results.
20. Noncardiac medical, psychiatric, and/or social disorder that would prevent successful completion of planned study testing or would invalidate its results.
21. Cardiac care, ongoing or planned, at a non-study center that would impede study completion.
22. For females: Pregnancy at the time of screening, pregnancy planned before study completion, or refusal to use an acceptable method of contraception for study duration if sexually active.
23. Unable to abstain or limit intake of grapefruit juice during the duration of the trial.
24. Refusal to provide written informed consent/assent.
25. In the opinion of the primary care physician, the subject is likely to be non-compliant with the study protocol.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Paridon, MD, Principal Investigator — Children's Hospital of Phildelphia
Locations (30):
- United States (26):
  - Phoenix Children's Hospital/Children's Heart Center at Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars/Sinai Heart Institute, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Cardiac Center/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Heart Institute, St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Hospital for Children/Herman B. Wells Center for Pediatric Research, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Congenital Heart Center/C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Mercy Hospital Kansas City, Kansas City, Missouri
  - Washington University St. Louis/St.Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska Children's Hospital and Medical Center, Omaha, Nebraska
  - Children's Hospital of New York, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hosptial, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Hospital/Dept. of Pediatric Cardiology, Salt Lake City, Utah
  - Seattle Children's Hosptial, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Stollery Children's Hospital - University of Alberta, Edmonton, Alberta
  - The Hospital for Sick Children, Toronto, Ontario
- South Korea (2):
  - Sejong General Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Children's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Maria MV, Goldberg DJ, Zak V, Hu C, Lubert AM, Dragulescu A, Mackie AS, McCrary A, Weingarten A, Parthiban A, Goot B, Goldstein BH, Taylor C, Lindblade C, Petit CJ, Spurney C, Harrild DM, Urbina EM, Schuchardt E, Beom Kim G, Kyoung Yoon J, Colombo JN, Files MD, Schoessling M, Ermis P, Wong PC, Garg R, Swanson SK, Menon SC, Srivastava S, Thorsson T, Johnson TR, Krishnan US, Paridon SM, Frommelt PC; Pediatric Heart Network. Impact of Udenafil on Echocardiographic Indices of Single Ventricle Size and Function in FUEL Study Participants. Circ Cardiovasc Imaging. 2022 Nov;15(11):e013676. doi: 10.1161/CIRCIMAGING.121.013676. Epub 2022 Nov 15. PMID 36378780
- [Derived] Goldberg DJ, Zak V, Goldstein BH, Schumacher KR, Rhodes J, Penny DJ, Petit CJ, Ginde S, Menon SC, Kim SH, Kim GB, Nowlen TT, DiMaria MV, Frischhertz BP, Wagner JB, McHugh KE, McCrindle BW, Shillingford AJ, Sabati AA, Yetman AT, John AS, Richmond ME, Files MD, Payne RM, Mackie AS, Davis CK, Shahanavaz S, Hill KD, Garg R, Jacobs JP, Hamstra MS, Woyciechowski S, Rathge KA, McBride MG, Frommelt PC, Russell MW, Urbina EM, Yeager JL, Pemberton VL, Stylianou MP, Pearson GD, Paridon SM; Pediatric Heart Network Investigators. Results of the FUEL Trial. Circulation. 2020 Feb 25;141(8):641-651. doi: 10.1161/CIRCULATIONAHA.119.044352. Epub 2019 Nov 17. PMID 31736357
- [Derived] Goldberg DJ, Zak V, Goldstein BH, McCrindle BW, Menon SC, Schumacher KR, Payne RM, Rhodes J, McHugh KE, Penny DJ, Trachtenberg F, Hamstra MS, Richmond ME, Frommelt PC, Files MD, Yeager JL, Pemberton VL, Stylianou MP, Pearson GD, Paridon SM; Pediatric Heart Network Investigators. Design and rationale of the Fontan Udenafil Exercise Longitudinal (FUEL) trial. Am Heart J. 2018 Jul;201:1-8. doi: 10.1016/j.ahj.2018.03.015. Epub 2018 Apr 3. PMID 29910047

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug | Placebo
Started | 200 | 200
Completed | 188 | 194
Not Completed | 12 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 7 | 4
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug | Placebo | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (2.033) | 15.6 (1.978) | 15.5 (2.005)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 72 | 161
  Male | 111 | 128 | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 25 | 56
  Not Hispanic or Latino | 168 | 174 | 342
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 21 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 13 | 23
  White | 169 | 155 | 324
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 2 | 9 | 11
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 11 | 19
  South Korea | 14 | 19 | 33
  United States | 178 | 170 | 348
Peak VO2 [Mean (Standard Deviation); unit: mL/kg/min] — The maximal rate of oxygen consumption during physical exertion as measured by a standardized exercise stress test protocol. These values were determined by clinical exercise physiologists at each of the participating centers after standardized training from the study team.
  mL/kg/min | 27.84 (6.877) | 28.01 (6.128) | 27.92 (6.50)
Weight [Mean (Standard Deviation); unit: kg] | 57.1 (13.925) | 59.0 (13.187) | 58.1 (13.577)
Maximal V02 at ventilatory anaerobic threshold (VAT) [Mean (Standard Deviation); unit: mL/kig/min] — The maximum rate of oxygen consumption at the VAT, defined as the point during exercise at which oxygen consumption is supplemented by anaerobic mechanisms. Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  mL/kig/min
    number analyzed (Participants) | 170 | 181 | 351
    (all) | 18.35 (4.633) | 17.71 (4.304) | 18.02 (4.471)
Ventilatory equivalents of carbon dioxide (VE/VCO2) at VAT [Mean (Standard Deviation); unit: Ratio] — This measure is a ratio of the amount of inspired air required to clear a given volume of CO2 from the circulation at the ventilatory anaerobic threshold (VAT). This measurement is made during exercise stress testing. Decreases in this ratio may reflect an improvement in ventilatory efficiency or an improvement in cardiac function. Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Ratio
    number analyzed (Participants) | 170 | 181 | 351
    (all) | 34.32 (4.845) | 34.75 (5.157) | 34.54 (5.006)
Respiratory rate at maximal exercise effort [Mean (Standard Deviation); unit: Breaths per minute] — The number of breaths taken per minute at maximum exercise effort. Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Breaths per minute
    number analyzed (Participants) | 199 | 200 | 399
    (all) | 51.11 (11.257) | 51.35 (12.676) | 51.23 (11.975)
Minute ventilation at maximal exercise effort [Mean (Standard Deviation); unit: L/min] — The amount of air inhaled or exhaled from the lungs per minute at maximal exercise effort. Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  L/min
    number analyzed (Participants) | 199 | 200 | 399
    (all) | 70.65 (21.055) | 75.84 (22.323) | 73.25 (21.828)
Work rate at maximal exercise effort [Mean (Standard Deviation); unit: Watts] — Work rate at the maximal exercise effort Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Watts
    number analyzed (Participants) | 198 | 199 | 397
    (all) | 119.68 (32.176) | 123.11 (32.140) | 121.40 (32.163)
Work rate at ventilatory anaerobic threshold (VAT) [Mean (Standard Deviation); unit: Watts] — Work rate at the VAT Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Watts
    number analyzed (Participants) | 167 | 177 | 344
    (all) | 66.19 (26.321) | 66.10 (23.446) | 66.14 (24.847)
Myocardial Performance Index (MPI) [Mean (Standard Deviation); unit: Ratio] — The MPI is a measure of systolic and diastolic function determined by velocities from blood pool Doppler assessment of the inflow and outflow tract of the dominant ventricle. MPI is calculated by dividing the sum of the isovolumetric contraction and relaxation time by the ejection time at each site measurement. The MPI is used to measure global cardiac dysfunction; decreases in MPI correspond with improved cardiac function and increases in MPI correspond with diminished cardiac function. The mean MPI in healthy people without heart disease is approximately 0.35. Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Ratio
    number analyzed (Participants) | 150 | 155 | 305
    (all) | 0.45 (0.172) | 0.45 (0.154) | 0.45 (0.163)
Log-transformed Reactive Hyperemia Index (lnRHI) [Mean (Standard Deviation); unit: Natural log-transformed RHI (lnRHI)] — Endothelial pulse amplitude tonometry (Endo-PAT) is a technique for the non-invasive assessment of peripheral vascular function. In adults, Endo-PAT has been demonstrated to identify those with coronary artery dysfunction and to correlate with brachial artery reactivity testing. Endo-PAT use in children has been more limited, but has shown excellent reproducibility. Reactive hyperemia index, a measure of the hyperemic response adjusted for baseline blood flow, is a measure of vascular function. A higher value denotes better, or more healthy, vascular (endothelial) function. Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Natural log-transformed RHI (lnRHI)
    number analyzed (Participants) | 191 | 192 | 383
    (all) | 0.46 (0.250) | 0.46 (0.332) | 0.46 (0.2936)
Log-transformed B-type natriuretic peptide (BNP) [Mean (Standard Deviation); unit: log(pg/mL)] — BNP is a hormone produced when the heart is enlarged or has to work harder to pump blood to the body. Higher BNP levels can be a sign of heart failure.
  BNP measurements reported as <2.0 were imputed as 1.0. Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  log(pg/mL)
    number analyzed (Participants) | 200 | 199 | 399
    (all) | 2.45 (1.003) | 2.26 (1.140) | 2.36 (1.076)
Pediatric Quality of Life Inventory (PedsQL) General Core Scale-Physical Functioning-Child reported [Mean (Standard Deviation); unit: Scores on a scale] — The PedsQL is a short questionnaire that has been used in multiple studies, including a previous study of Fontan patients. Total scores were calculated using the Scoring Dimensions Calculation described under PedsQL TM 4.0 Generic Core Scales. In general, higher scores correspond with perceived improvement in quality of life (QoL). Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Scores on a scale
    number analyzed (Participants) | 196 | 200 | 396
    (all) | 72.52 (16.805) | 73.35 (16.686) | 72.94 (16.729)
PedsQL General Core Scale-Physical Functioning-Parent reported [Mean (Standard Deviation); unit: Scores on a scale] — The PedsQL is a short questionnaire that has been used in multiple studies, including a previous study of Fontan patients. Total scores were calculated using the Scoring dimensions calculation described under PedsQL TM 4.0 Generic Core Scales section. Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Scores on a scale
    number analyzed (Participants) | 194 | 193 | 387
    (all) | 71.58 (18.155) | 73.18 (18.006) | 72.38 (18.075)
PedsQL General Core Scale-Psychosocial Health Summary Score-Child reported [Mean (Standard Deviation); unit: Scores on a scale] — Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Scores on a scale
    number analyzed (Participants) | 196 | 200 | 396
    (all) | 71.90 (16.976) | 72.30 (16.811) | 72.10 (16.872)
PedsQL General Core Scale-Psychosocial Health Summary Score-Parent reported [Mean (Standard Deviation); unit: Scores on a scale] — Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Scores on a scale
    number analyzed (Participants) | 194 | 193 | 387
    (all) | 68.48 (16.130) | 70.51 (17.525) | 69.49 (16.849)
PedsQL Cardiac Module Scale-Treatment II [Mean (Standard Deviation); unit: Scores on a scale] — Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Scores on a scale
    number analyzed (Participants) | 178 | 185 | 363
    (all) | 87.84 (9.769) | 89.35 (9.288) | 88.61 (9.544)
PedsQL Cardiac Module Scale-Perceived Physical Appearance [Mean (Standard Deviation); unit: Scores on a scale] — Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Scores on a scale
    number analyzed (Participants) | 195 | 200 | 395
    (all) | 74.23 (24.291) | 75.92 (25.185) | 75.09 (24.731)
PedsQL Cardiac Module Scale-Treatment Anxiety [Mean (Standard Deviation); unit: Scores on a scale] — Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Scores on a scale
    number analyzed (Participants) | 194 | 200 | 394
    (all) | 79.99 (23.164) | 80.09 (23.736) | 80.04 (23.426)
PedsQL Cardiac Module Scale-Cognitive Problems [Mean (Standard Deviation); unit: Scores on a scale] — Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Scores on a scale
    number analyzed (Participants) | 195 | 198 | 393
    (all) | 64.67 (20.709) | 65.23 (22.967) | 64.95 (21.850)
PedsQL Cardiac Module Scale-Communication Problems [Mean (Standard Deviation); unit: Scores on a scale] — Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment.
  Scores on a scale
    number analyzed (Participants) | 195 | 199 | 394
    (all) | 74.74 (21.933) | 72.63 (22.938) | 73.67 (22.443)
Pediatric Cardiac Quality of Life Inventory (PCQLI) Total Score-Ages 8 to 12-Child reported [Mean (Standard Deviation); unit: Scores on a scale] — The PCQLI is a disease-specific assessment of health-related quality of life for children or adolescents with congenital or acquired heart disease. Total scores were calculated using the Total Scores calculationwhich is a composite of multiple subscales (disease impact, emotional functioning, and communication). The Total Score is derived by summing individual subscale scores and converting them to a scale ranging from 0 to 100. Higher scores correspond with perceived improvement in quality of life (QoL). Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment. Only participants aged 8 to 12 were included in this assessment.
  Scores on a scale
    number analyzed (Participants) | 28 | 19 | 47
    (all) | 69.04 (15.091) | 75.55 (14.392) | 71.67 (15.005)
PCQLI Total Score-Ages 8 to 12-Parent reported [Mean (Standard Deviation); unit: Scores on a scale] — The PCQLI is a disease-specific assessment of health-related quality of life for children or adolescents with congenital or acquired heart disease. Total scores were calculated using the Total Scores calculation and was derived by summing individual subscale scores (disease impact, emotional functioning, and communication) and converting them to a scale ranging from 0 to 100. In general, higher scores correspond with perceived improvement in quality of life (QoL). Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment. Only parents with participants aged 8 to 12 were included in this assessment.
  Scores on a scale
    number analyzed (Participants) | 29 | 18 | 47
    (all) | 65.56 (18.078) | 70.27 (16.809) | 67.36 (17.570)
PCQLI Total Score-Ages 13 to 18-Child reported [Mean (Standard Deviation); unit: Scores on a scale] — The PCQLI is a disease-specific assessment of health-related quality of life for children or adolescents with congenital or acquired heart disease. Total scores were calculated using the Total Scores calculation. In general, higher scores correspond with perceived improvement in quality of life (QoL). Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment. Only participants aged 13 to 18 were included in this assessment.
  Scores on a scale
    number analyzed (Participants) | 167 | 179 | 346
    (all) | 73.39 (14.979) | 73.62 (14.790) | 73.51 (14.860)
PCQLI Total Score-Ages 13 to 18-Parent reported [Mean (Standard Deviation); unit: Scores on a scale] — The PCQLI is a disease-specific assessment of health-related quality of life for children or adolescents with congenital or acquired heart disease. Total scores were calculated using the Total Scores calculation. In general, higher scores correspond with perceived improvement in quality of life (QoL). Population: Not all participants had a Baseline value due to errors in data capture and/or the participant did not complete the assessment. Only parents of participants aged 13 to 18 were included in this assessment.
  Scores on a scale
    number analyzed (Participants) | 163 | 177 | 340
    (all) | 70.23 (15.001) | 72.74 (15.970) | 71.54 (15.541)

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximal VO2 From Baseline to Week 26 Using Last Observation Carried Forward (LOCF)
Description: The change in exercise capacity (as measured by peak VO2 at maximum exercise effort) from baseline to 26 weeks
Time Frame: Baseline to 26 Weeks
Population: Intent to Treat Population
Measure: Mean (Standard Deviation); unit: mL/kg/min
Groups:
- Udenafil: Intent to Treat Population on active drug.
- Placebo: Intent to Treat Population on Placebo
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 200 | 200
mL/kg/min | -0.23 (4.056) | -0.89 (3.672)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; It was estimated that a sample size of 198 participants per group would provide 90% power to detect a mean treatment group difference in change from baseline to Week 26 in maximal VO2 scores of 10% (ie, an improvement of 2.8 mL/kg/min in the udenafil group compared to 0 in the control group, assuming a Type I error of 0.05 and standard deviation of 7.235). A difference of 2.8, equivalent to a 10% increase from a baseline of 28 mL/kg/min, represents approximately 0.4 standard deviations; Test type: Superiority; p = 0.092, ANCOVA — LS mean was the estimated treatment difference from the analysis model; ANCOVA fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline maximal VO2. LOCF imputation used; Mean Difference (Final Values) = 0.64, Standard Error of Mean 0.377

2. Secondary Outcome: Change in Myocardial Performance Index (MPI) From Baseline to Week 26
Description: Change in the myocardial performance index (MPI) from baseline to 26 weeks is determined by velocities from blood pool Doppler of the inflow and outflow tract of the dominant ventricle. The measure is the ratio of the sum of isovolumetric contraction time and isovolumetric relaxation time, divided by ventricular ejection time. A lower value is consistent with a more efficient ventricle (better function). A value of zero indicates that there is no isovolumetric contraction or relaxation and, while physiologically implausible, would be consistent with a perfectly efficient ventricle. The mean left ventricular MPI in healthy people without heart disease is approximately 0.35 while the mean right ventricular MPI is approximately 0.1 due to the reduced ventricular afterload of the pulmonary circulation. In general, a decrease in the MPI corresponds to more efficient (better) ventricular function, while an increase in MPI corresponds to less efficient (worse) ventricular function.
Time Frame: Week 26
Population: This analysis was performed only on participants with paired data. For variety of technical reasons the quality of echocardiographic images were not sufficient to allow for accurate assessment of the MPI in a subset of participants. These reasons include poor acoustic windows and noisy Doppler signal.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 122 | 128
ratio | -0.02 (0.112) | 0.01 (0.132)
Statistical Analysis 1: Comparison: Drug vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.024, ANCOVA — LS mean was the estimated treatment difference from the analytical model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline maximal VO2; Mean Difference (Final Values) = -0.03, Standard Error of Mean 0.014

3. Secondary Outcome: Change in Log-transformed Reactive Hyperemia Index (InRH) From Baseline to Week 26
Description: Endothelial pulse amplitude tonometry (Endo-PAT) is a technique for the non-invasive assessment of peripheral vascular function. In adults, Endo-PAT has been demonstrated to identify those with coronary artery dysfunction and to correlate with brachial artery reactivity testing. Endo-PAT use in children has been more limited, but has shown excellent reproducibility. Reactive hyperemia index, a measure of the hyperemic response adjusted for baseline blood flow, is a measure of vascular function. A higher value denotes better, or more healthy, vascular (endothelial) function.
Time Frame: Week 26
Population: This analysis was performed only on participants with paired data. For variety of technical reasons the signal for the reactive hyperemia index was not sufficient to allow for accurate assessment of the index in a subset of participants.
Measure: Mean (Standard Deviation); unit: Natural log-transformed RHI (lnRHI)
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 175 | 184
Natural log-transformed RHI (lnRHI) | 0.06 (0.301) | 0.04 (0.364)
Statistical Analysis 1: Comparison: Drug vs Placebo; Test type: Superiority; p = 0.591, ANCOVA; Mean Difference (Final Values) = 0.02, Standard Error of Mean 0.591

4. Secondary Outcome: Change in Serum Brain-type Natriuretic Peptide (BNP) From Baseline to Week 26.
Description: BNP is a hormone produced when the heart is enlarged or has to work harder to pump blood to the body. Higher levels of BNP can be a sign of heart failure.
Time Frame: Week 26
Population: This analysis was performed on a subset of patients who had analyzable lab samples at both baseline and 26 weeks.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 187 | 191
pg/mL | 0.08 (0.905) | 0.03 (1.137)
Statistical Analysis 1: Comparison: Drug vs Placebo; Test type: Superiority; p = 0.169, ANCOVA; Mean Difference (Final Values) = 0.13, Standard Error of Mean 0.094

5. Secondary Outcome: Change in VO2 at VAT
Description: This outcome measures the change in milliliters of oxygen consumption (VO2) per minute at the ventilatory anaerobic threshold (VAT) between Week 26 and Baseline Visits using last observation carried forward (ITT Population). The anaerobic threshold is the period in exercise when metabolism switches from aerobic to anaerobic. This is an useful measure of submaximal exercise capacity particularly in the single ventricle population.
Time Frame: 26 Weeks
Population: Data from the anaerobic threshold is not calculable for all participants given noise within the data tracings. These data are from the intent to treat (ITT) analyses for all participants for whom a baseline value was calculable.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 170 | 181
mL/kg/min | -0.07 (2.998) | -0.68 (3.216)
Statistical Analysis 1: Comparison: Drug vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.012, ANCOVA — LS mean was the estimated treatment mean difference from the analysis model; Fixed factors: ventricular morphology and treatment group, with a continuous covariate of Baseline maximal VO2. LOCF imputation; Median Difference (Final Values) = 0.78, Standard Error of Mean 0.308

6. Secondary Outcome: Change in Work Rate at VAT From Baseline to Week 26 With LOCF
Description: This outcome measures the change in work (measured in Watts) at the ventilatory anaerobic threshold (VAT) between Week 26 and Baseline Visits using last observation carried forward (ITT Population). The anaerobic threshold is the period in exercise when metabolism switches from aerobic to anaerobic. This is an useful measure of submaximal exercise capacity particularly in the single ventricle population.
Time Frame: 26 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 167 | 177
Watts | 3.46 (15.076) | 0.31 (13.246)
Statistical Analysis 1: Comparison: Drug vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.029, ANCOVA — LS mean was the estimated treatment difference in the analysis model; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 3.20, Standard Error of Mean 1.460

7. Secondary Outcome: Change in VE/VCO2 at VAT From Baseline to Week 26
Description: This measure is a ratio of the amount of inspired air required to clear a given volume of CO2 from the circulation at the ventilatory anaerobic threshold (VAT). This measurement is made during exercise stress testing. Decreases in this ratio may reflect an improvement in ventilatory efficiency or an improvement in cardiac function.
Time Frame: 26 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 170 | 181
Ratio | -0.76 (3.564) | -0.05 (2.967)
Statistical Analysis 1: Comparison: Drug vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.011, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline maximal VO2. LOCF imputation; Mean Difference (Final Values) = -0.82, Standard Error of Mean 0.321

8. Secondary Outcome: Change in Respiratory Rate at Maximal Exercise Effort From Baseline to Week 26 Using LOCF
Time Frame: Week 26
Population: ITT Population. Of note, some participants may not have had Baseline values due to errors in data capture and/or the participant did not complete the assessment, but was encouraged to come back to complete Week 26 assessments. Only participants with both a Baseline value and a Week 26 value were included in the analysis.
Measure: Mean (Standard Deviation); unit: Breaths/min
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 199 | 200
Breaths/min | -1.01 (10.030) | -1.44 (9.928)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.696, ANCOVA; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline VO2. LOCF imputation; Mean Difference (Final Values) = 0.35, Standard Error of Mean 0.903

9. Secondary Outcome: Change in Minute Oxygen Consumption at Maximal Exercise Effort From Baseline to Week 26
Description: The amount of air that enters the lungs per minute at maximal exercise effort.
Time Frame: Week 26
Population: ITT Population. Of note, some participants may not have had baseline values due to errors in data capture and/or not completing the assessment, but were encouraged to come back to complete Week 26 assessments. Only participants with both a baseline value and a Week 26 value were included in the analysis.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 199 | 200
L/min | 1.15 (13.934) | -0.10 (13.748)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.915, ANCOVA — LS mean was the estimated treatment difference from the analysis model; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.14, Standard Error of Mean 1.319

10. Secondary Outcome: Change in Work Rate at Maximal Exercise Effort Between Baseline and Week 26 Using LOCF
Description: Change in power at maximal exercise effort.
Time Frame: Week 26
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Watts
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 198 | 199
Watts | 2.99 (14.334) | 2.45 (13.503)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; LS mean differences between treatment groups were analyzed; Test type: Superiority; p = 0.891, ANCOVA — LS mean was the estimated treatment difference from the analysis model; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = 0.19, Standard Error of Mean 1.363

11. Secondary Outcome: Change in Pediatric Quality of Life (PedsQL) Generic Core Scales - Physical Functioning Subscale (Child Reported)
Description: The PedsQL is a short questionnaire that has been used in multiple studies, including a previous study of Fontan patients. A 5-point Likert response scale (0-4) is used. This score was linearly transformed on a scale of 0-100 (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0). For an individual, a higher score is associated with a higher reported healthcare-related quality of life. For each population (treatment and placebo), population means were calculated at baseline and 26 weeks. The outcome measure is the difference between week 26 and baseline (week 26 - baseline).
Time Frame: 26 weeks
Population: ITT Population. Of note, some participants may not have had Baseline values due to errors in data capture and/or not completing the assessment, but were encouraged to come back and complete the Week 26 assessments. Only participants with both a Baseline and a Week 26 value were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 186 | 193
Scores on a scale | 2.08 (12.006) | 1.53 (11.823)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.691, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group, with a continuous covariate of Baseline physical functioning (child reported); Mean Difference (Final Values) = 0.44, Standard Error of Mean 1.100

12. Secondary Outcome: Change in Pediatric Quality of Life (PedsQL) Generic Core Scales - Physical Functioning Subscale (Parent Reported)
Description: as for outcome 11
Time Frame: 26 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 181 | 181
Scores on a scale | 2.74 (18.011) | 1.94 (15.328)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.985, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline physical functioning (parent reported); Mean Difference (Final Values) = 0.03, Standard Error of Mean 1.544

13. Secondary Outcome: Change in Pediatric Quality of Life (PedsQL) Generic Core Scales - Psychosocial Health Subscale (Child Reported)
Description: as for outcome 11
Time Frame: 26 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 185 | 193
Scores on a scale | 2.84 (11.356) | 1.74 (10.700)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.273, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline psychosocial health summary score (child reported); Mean Difference (Final Values) = 1.14, Standard Error of Mean 1.039

14. Secondary Outcome: Change in Pediatric Quality of Life (PedsQL) Generic Core Scales - Psychosocial Health Subscale (Parent Reported)
Description: as for outcome 11
Time Frame: 26 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 181 | 181
Scores on a scale | 2.64 (13.546) | 2.15 (13.737)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.966, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline psychosocial health summary score (parent reported); Mean Difference (Final Values) = -0.06, Standard Error of Mean 1.327

15. Secondary Outcome: Change in Pediatric Quality of Life (PedsQL) Inventory - Cardiac Module Scale - Treatment II Subscale (Child-reported)
Description: as for outcome 11
Time Frame: 26 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 164 | 173
Scores on a scale | 0.24 (11.655) | -0.09 (9.046)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.706, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline cardiac module scale (Treatment II); Mean Difference (Final Values) = -0.38, Standard Error of Mean 1.011

16. Secondary Outcome: Change in Pediatric Quality of Life (PedsQL) Inventory - Cardiac Module Scale - Perceived Physical Appearance Subscale
Description: as for outcome 11
Time Frame: 26 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 184 | 192
Scores on a scale | 2.45 (20.819) | 0.78 (17.396)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.382, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline cardiac module scale (perceived physical appearance); Mean Difference (Final Values) = 1.50, Standard Error of Mean 1.707

17. Secondary Outcome: Change in Pediatric Quality of Life (PedsQL) Inventory - Cardiac Module Scale - Treatment Anxiety Subscale
Description: as for outcome 11
Time Frame: 26 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 184 | 192
Scores on a scale | 3.37 (19.258) | 1.66 (16.477)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.236, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline cardiac module scale (treatment anxiety); Mean Difference (Final Values) = 1.91, Standard Error of Mean 1.611

18. Secondary Outcome: Change in Pediatric Quality of Life (PedsQL) Inventory - Cardiac Module Scale - Cognitive Problems Subscale
Description: as for outcome 11
Time Frame: 26 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 183 | 192
Scores on a scale | 2.19 (16.826) | 3.05 (17.027)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.543, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline cardiac module scale (cognitive problems); Mean Difference (Final Values) = -0.99, Standard Error of Mean 1.622

19. Secondary Outcome: Change in Pediatric Quality of Life (PedsQL) Inventory - Cardiac Module Scale - Communication Problems Subscale
Description: The PedsQL is a short questionnaire that has been used in multiple studies, including a previous study of Fontan patients. A 5-point Likert response scale (0-4) is used. This score was linearly transformed on a scale of 0-100 (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0). For an individual, a higher score is associated with a higher reported healthcare-related quality of life. For each population (treatment and placebo), population means were calculated at baseline and 26 week. The outcome measure is the difference between week 26 and baseline (week 26 - baseline).
Time Frame: 26 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 183 | 192
Scores on a scale | 1.82 (20.406) | 4.36 (17.954)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.352, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline cardiac module scale (communication problems); Mean Difference (Final Values) = -1.66, Standard Error of Mean 1.780

20. Secondary Outcome: Change in Pediatric Cardiac Quality of Life Inventory (PCQLI) Total Score-Ages 8 to 12 (Child Reported)
Description: The PCLQI is a disease-specific measure of health-related quality of life for children and adolescents with congenital or acquired heart disease. The PCQLI score is calculated by adding together the scores from the two subscales: Disease Impact and Psychosocial Impact. Each subscale can score a maximum of 50 points, resulting in a total score with a maximum of 100. Higher scores indicate better perceived health-related quality of life. For each population (treatment and placebo), population means were calculated at baseline and 26 weeks. The outcome measure is the difference between week 26 and baseline (week 26 - baseline).
Time Frame: 26 weeks
Population: ITT Population. Of note, some participants may not have had Baseline values due to errors in data capture and/or not completing the assessment, but were encouraged to come back and complete the Week 26 assessments. Only participants with both a Baseline and a Week 26 value who were aged 8 to 12 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 16 | 12
Scores on a scale | 3.26 (12.287) | -2.37 (16.368)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.533, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors of ventricular morphology and treatment group with a continuous covariate of Baseline total score (age 8-12, child reported); Mean Difference (Final Values) = 3.59, Standard Error of Mean 5.684

21. Secondary Outcome: Change in Pediatric Cardiac Quality of Life Inventory (PCQLI) Total Score-Ages 8 to 12 (Parent Reported)
Description: as for outcome 20
Time Frame: 26 weeks
Population: ITT Population. Of note, some participants may not have had Baseline values due to errors in data capture and/or not completing the assessment, but were encouraged to come back and complete the Week 26 assessments. Only participants with both a Baseline and a Week 26 value were included in the analysis. Only parents with participants aged 8-12 were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 17 | 11
Scores on a scale | -0.91 (13.399) | -4.44 (6.389)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.654, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline total score (age 8-12, parent reported); Mean Difference (Final Values) = 1.84, Standard Error of Mean 4.057

22. Secondary Outcome: Change in Pediatric Cardiac Quality of Life Inventory (PCQLI) Total Score-Ages 13 to 18 (Child Reported)
Description: as for outcome 20
Time Frame: 26 weeks
Population: ITT Population. Of note, some participants may not have had Baseline values due to errors in data capture and/or not completing the assessment, but were encouraged to come back and complete the Week 26 assessments. Only participants aged 13-18 with both a Baseline and a Week 26 value were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 158 | 170
Scores on a scale | -0.08 (11.032) | 0.09 (9.626)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment groups were analyzed; p = 0.963, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors: ventricular morphology and treatment group with a continuous covariate of Baseline total score (ages 13-18, child reported); Mean Difference (Final Values) = -0.05, Standard Error of Mean 1.069

23. Secondary Outcome: Change in Pediatric Cardiac Quality of Life Inventory (PCQLI) Total Score-Ages 13 to 18 (Parent Reported)
Description: as for outcome 20
Time Frame: 26 weeks
Population: ITT Population. Of note, some participants may not have had Baseline values due to errors in data capture and/or not completing the assessment, but were encouraged to come back and complete the Week 26 assessments. Only parents of participants aged 13-18 with both a Baseline and a Week 26 value were included in the analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Udenafil | Placebo
Number analyzed (Participants) | 152 | 162
Scores on a scale | 0.36 (11.722) | -1.60 (11.179)
Statistical Analysis 1: Comparison: Udenafil vs Placebo; Test type: Superiority — LS mean differences between treatment group were analyzed; p = 0.246, ANCOVA — LS mean was the estimated treatment difference from the analysis model; Fixed factors of ventricular morphology and treatment group with a continuous covariate of Baseline total score (ages 13-18, parent reported); Mean Difference (Final Values) = 1.36, Standard Error of Mean 1.171

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded over the 26 weeks of study period plus an additional 3 months of follow-up.
Arm/Group | Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/200
Serious Adverse Events (participants affected / at risk) | 14/200 | 10/200
Other Adverse Events (participants affected / at risk) | 158/200 | 135/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug (N=200) | Placebo (N=200)
Retinal Artery Thrombosis (Eye disorders) | 1 (1) | 0 (0) — Central retinal artery and vein occlusion of unclear etiology was confirmed with fluorescein angiogram
Diplegia (Nervous system disorders) | 1 (1) | 0 (0) — Subject described a tingly, pins and needles feeling on his legs, his gait was unstable, and he experienced an episode of urinary incontinence
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) — Shortness of breath, shortness of breath on exertion, and tightness of chest.
Palpitation (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) — Fainted
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Gastrointestinal hemorhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Protein-losing gastroenteropathy (Endocrine disorders) | 1 (2) | 0 (0)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Arrthythema (Vascular disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Bipolar I disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Intracardiac Thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cerebral Vascular Accident (Vascular disorders) | 0 (0) | 1 (1)
Fatigue (Nervous system disorders) | 0 (0) | 1 (1)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infections (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug (N=200) | Placebo (N=200)
Nausea (Gastrointestinal disorders) | 16 (200) | 9 (200)
Vomiting (Gastrointestinal disorders) | 15 (200) | 5 (200)
Chest Pain (General disorders) | 9 (200) | 16 (200)
Nasopharyngitis (Infections and infestations) | 13 (200) | 9 (200)
Upper Respiratory Tract Infectins (Infections and infestations) | 24 (200) | 22 (200)
Dizziness (Nervous system disorders) | 16 (200) | 17 (200)
Headache (Nervous system disorders) | 79 (200) | 51 (200)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 (200) | 5 (200)
Flushing (Vascular disorders) | 32 (200) | 12 (200)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-27): https://cdn.clinicaltrials.gov/large-docs/15/NCT02741115/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT02741115/SAP_001.pdf